CLINICAL TRIAL: NCT00327379
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Design, 2-Arm Study to Investigate the Effect of Aprotinin on Transfusion Requirements in Patients Undergoing Elective Spinal Fusion Surgery
Brief Title: Effect of Aprotinin on Transfusion Requirements in Patients Undergoing Elective Spinal Fusion Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11799; 2005-003999-38 (EudraCT Number)
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Blood Loss, Surgical; Postoperative Hemorrhage
Keywords: Bloodloss; Transfusion Requirements in Patients Undergoing Elective Spinal Fusion Surgery
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage | interventions — Aprotinin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Trasylol (Aprotinin, BAYA0128)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trasylol (Aprotinin, BAYA0128) — Infusion of aprotinin (loading dose of 2 million KIU (Kallikrein Inhibitor Units) followed by 500,000 KIU/hour until the end of surgery)
  Arms: Arm 1
Drug: Placebo — Infusion of placebo (loading dose of 2 million KIU (Kallikrein Inhibitor Units) followed by 500,000 KIU/hour until the end of surgery)
  Arms: Arm 2

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of aprotinin as compared to placebo, in reducing the need for blood transfusion in adult subjects undergoing elective spinal fusion surgery involving 3 to 7 vertebral levels with instrumentation

ELIGIBILITY:
Inclusion Criteria:

* Subjects requiring elective spinal fusion surgery involving 3 to 7 vertebral levels with instrumentation. One vertebral level is defined as encompassing two vertebral bodies and one inter-vertebral disc space, so that a contiguous spinal fusion involving 3 vertebral levels would include 4 vertebral bodies and 3 inter-vertebral disc spaces.

Exclusion Criteria:

* Subjects with previous exposure to aprotinin in the last 6 months. If the subject has undergone cardiac surgery in the last 6 months, all attempts should be made to ascertain if aprotinin was administered during cardiac surgery. If no records are available, or if the subject received aprotinin, the subject should be excluded.- Subjects with a known or suspected allergy to aprotinin.
* Subjects with sepsis or a known bone infection.- Subjects with known bone malignancy.
* Subjects with a creatinine clearance less than 30mL/min as calculated by the Cockcroft-Gault formula.
* Subjects with a history of bleeding diathesis or known coagulation factor deficiency.
* Subjects with failure of a major organ system or any active significant medical illness that in the opinion of the Investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study
* Subjects who refuse to receive allogenic blood products for religious or other reasons.
* Subjects whose preoperative red blood cell volume is so low that a blood transfusion would be likely to be given perioperatively (preoperative hematocrit or hemoglobin values <24% or <8 g/dl, respectively).
* Subjects who have participated in an investigational drug study within the past 30 days
* Subjects with a history of deep vein thrombosis or pulmonary embolism.
* Subjects who are pregnant or breast feeding.
* Women of childbearing potential in whom the possibility of pregnancy cannot be excluded by a negative serum pregnancy test at screening.
* Women of childbearing potential who are not using a reliable method of contraception.
* Planned use of other antifibrinolytic agents.
* Subjects on chronic anticoagulant treatment with Vit K antagonists that cannot be temporarily discontinued for the surgical procedure (as per local practices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-02-27 (Actual); Primary Completion 2007-03-01 (Actual); Study Completion 2007-03-01 (Actual)

PRIMARY OUTCOMES:
Percent of patients requiring a blood transfusion (blood or packed red blood cells, autologous or allogenic) | anytime in the intra-operative or postoperative period (up to the earlier of Day 7 or discharge).

SECONDARY OUTCOMES:
The percent of patients receiving an allogenic transfusion of blood or packed red cells during surgery and up to the earlier of Day 7 or discharge | surgery to discharge
The percent of patients who did and did not predonate blood receiving an allogenic transfusion of blood or packed red cells during surgery and up to the earlier of Day 7 or discharge | surgery to discharge
The number of units of blood or packed red cells transfused. There will be analyses for the combination of autologous and allogenic transfusion and for allogenic alone | surgery to discharge
The number of units of blood or packed red cells transfused per patient requiring transfusion | surgery to discharge
Drainage (in milliliters) from the operative site in the first 8 hours postoperatively, and total drainage until removal of drains or until hospital discharge (whichever is earlier) | surgery to discharge
Blood loss during surgery, based on qualitative and quantitative estimates | surgery
The change from preoperative hemoglobin concentration to postoperative hemoglobin concentration (obtained in the morning of Day 3, or, if transfused earlier, prior to transfusion). | pre-op and day 3 post surgery
Surgeons assessment of the degree to which bleeding obscured his/her view of the surgical field, relative to past, similar procedures | surgery to discharge
The percent of patients receiving colloid or other blood products, and the number of units transfused | surgery to discharge
Changes in blood markers related to inflammation and blood coagulation | surgery to discharge
Changes in FEV1 | surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Canada (3):
  - Oshawa, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
- Germany (4):
  - Karlsbad, Baden-Wurttemberg
  - Münster, North Rhine-Westphalia
  - Neustadt, Schleswig-Holstein
  - Berlin
- Spain (4):
  - Barcelona
  - Madrid
  - Pamplona
  - Valencia

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/